CLINICAL TRIAL: NCT02493738
Title: A Phase I Single-Center, Randomized, Open-label, Single Dose, Crossover Study in Korean Healthy Male Volunteers to Evaluate Pharmacokinetics of Lozanoc and Sporanox
Brief Title: A Clinical Study to Evaluate the Pharmacokinetics of Lozanoc and Sporanox in Korean Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: BR-ITR-CT-101
Record Dates: First submitted 2015-07-07; First posted 2015-07-09 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: Superficial Mycoses; Dermatomycoses; Candidiasis; Histoplasmosis
MeSH Terms: conditions — Dermatomycoses; Candidiasis; Histoplasmosis | interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lozanoc 50mg (Experimental): Lozanoc 50mg, oral administration
  Interventions: Drug: Lozanoc 50mg
- Sporanox 100mg (Active Comparator): Sporanox 100mg, oral administration
  Interventions: Drug: Sporanox 100mg

INTERVENTIONS:
Drug: Lozanoc 50mg — Lozanoc 50mg single dose under fed and fasted condition
  Arms: Lozanoc 50mg
Drug: Sporanox 100mg — Sporanox 100mg single dose under fed condition
  Arms: Sporanox 100mg

SUMMARY:
Study Objectives:

* To evaluate the pharmacokinetics (PK) of orally administered Lozanoc under fasted and fed condition in healthy male subjects
* To compare the pharmacokinetics (PK) of orally administered Lozanoc and Sporanox under fed condition in healthy male subjects
* To evaluate the safety and tolerability of single oral dose of Lozanoc and Sporanox in Korean healthy male subjects

DETAILED DESCRIPTION:
Phase I Study divided into 3 parts written as bellows.

Part I. Lozanoc 50mg single dose under fed condition vs Part 2. Lozanoc 50mg single dose under fasted condition vs Part 3. Sporanox 100mg single dose under fed condition

ELIGIBILITY:
Inclusion Criteria:

1. Korean male volunteers in the age between 19 and 50 years old (inclusive)
2. Subject who are able to give signed informed consent
3. Body mass index (BMI) in the range of 19 to 28 kg/m2 and weighting at least 50kg
4. Subject who are considered

   * Pre-study physical examination with no clinically significant abnormalities
   * No clinically significant medical history
   * Vital signs were to be within reference ranges, or if outside of the range, not deemed clinically significant in the opinion of the Investigator

     * 90 mmHg ≤ systolic blood pressure (sitting position) ≤ 140mmHg
     * 50 mmHg ≤ diastolic blood pressure (sitting position) ≤ 90 mmHg
   * Pre-study clinical laboratory findings were to be within reference range, or if outside of the range, not deemed clinically significant in the opinion of the Investigator
   * No clinically significant abnormalities in 12-lead ECG results
5. Agree to continue to use at least two accepted methods of birth control and not to donate sperm for at least 1 days before the first dosing, during the course of the study and for a period of 90days following the last dosing.

   * Acceptable methods of birth control are: female (sexual partner) hormonal contraceptives; intrauterine device; surgical sterility at least 6 months prior to screening (Ex. hysterectomy, bilateral oophorectomy, and/or tubal ligation); use diaphragm; use condom; or spermicide

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

1. History of allergy or sensitivity to any drug, including any prior serious adverse reaction to antifungal agent(s)
2. History of congestive heart failure or Patients with ventricular dysfunction such as congestive heart failure
3. Undergone surgery or who have a medical condition, that in the judgment of the Investigator, may affect absorption, distribution, metabolism or elimination of the drug product
4. Participated in a previous clinical trial within 90 days prior to screening visit
5. Donated blood or had a significant loss of blood within 60 days prior to screening visit
6. Special diet or substantial changes in eating habits within 30 days prior to screening visit
7. Use of any prescription medication within 14 days before screening visit
8. Use of any other OTC medication within the 7 days before screening visit
9. History of smoking within 3 months prior to screening visit
10. Have a recent history (within 2 years prior to the screening visit) of alcohol or drug abuse or a positive screen for drugs of abuse at screening
11. Positive blood screen for HIV or hepatitis B or C or syphilis
12. Clinically important abnormal hepatic function test (AST, ALT greater than 2 fold of reference upper limit (ULN), or total bilirubin greater than 1.5 x ULN)
13. Not suitable to participate in the study in the opinion of the Investigator including an existing physical or mental condition that prevents compliance with the protocol

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Cmax | 0~120 hour after medication

SECONDARY OUTCOMES:
tmax | 0~120 hour after medication
AUCinf | 0~120 hour after medication

CONTACTS AND LOCATIONS:
Overall Officials: Kyun-Seop Bae, M.D., Ph.D., Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea